CLINICAL TRIAL: NCT00418977
Title: Early Identification and Treatment of Anorexia Nervosa
Brief Title: Comparing the Effectiveness of Two Therapies to Treat Signs of Anorexia Nervosa in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 04-0978; K23MH074506 (NIH); DSIR 84-CTS
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Eating Disorders
Keywords: Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Based Therapy (Experimental): Participants will receive family based therapy (FBT)
  Interventions: Behavioral: Family-Based Therapy ("Maudsley Method")
- Individual Supportive Psychotherapy (Active Comparator): Participants will receive individual supportive psychotherapy (ISP)
  Interventions: Behavioral: Individual Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Family-Based Therapy ("Maudsley Method") — The goal of FBT is to resolve the eating disorder and return the patient to healthy psychosocial and physiological development through active family involvement across three treatment phases. In Phase I, therapy is focused on the disordered eating. The therapist primarily makes careful, persistent requests for united parental action toward re-feeding and/or regulating eating habits and directs the discussion so as to create and reinforce a strong parental alliance around their efforts at feeding their child. In Phase II, the goal is to gradually transfer control over eating back to the participant, with the parents still maintaining general oversight and responsibility for continued progression toward healthy habits. In Phase III, the central goal is establishment of a healthy child or adolescent relationship with the parents where disordered eating is not the basis of interaction.
  Other Names: FBT; Maudsley Method
  Arms: Family Based Therapy
Behavioral: Individual Supportive Psychotherapy — The goal of ISP is for the patient to understand and address the psychological issues underlying the origin and maintenance of the eating disorder. This work is done directly with the child/adolescent. In this treatment, eating disorders are seen as complicated (e.g., they tend to mask other underlying difficulties). In Phase I, the aims are to establish a sound therapeutic relationship, obtain a comprehensive description of the eating problem and its development, identify underlying problems that might be responsible for the disordered eating, and inform the patient about the dangers of eating disorders. Phase II encourages participants to explore underlying emotional problems, facilitates self-disclosure and expression of feelings, and fosters independence. Phase III focuses on how other underlying issues might affect future adjustment.
  Other Names: ISP
  Arms: Individual Supportive Psychotherapy

SUMMARY:
This study will compare the effectiveness of two therapies to treat early signs of anorexia nervosa in adolescents.

DETAILED DESCRIPTION:
Eating disorders often result in serious illness and can lead to prolonged health complications, including heart and kidney problems, digestive disorders, nerve damage, and low blood pressure. Anorexia nervosa is a type of eating disorder in which a person does not eat enough for fear of becoming overweight, resulting in extreme weight loss. Women are at a greater risk of developing this disease, particularly when they are between the ages of 12 and 24. Treatments for anorexia nervosa typically include nutrition counseling, psychotherapy, and medication. The purpose of this study is to compare the effectiveness of two therapies to treat adolescents who have signs of anorexia nervosa but have not fully developed the disease.

Potential participants will attend 2 screening visits during which parents and children will complete separate questionnaires and undergo 3 interviews regarding eating behaviors and changes in mood. Once screening evaluations have been completed, eligible participants will be randomly assigned to 1 of 2 treatment groups. Participants assigned to the first group will receive 14 family therapy sessions. All family members living with the child will be asked to attend these sessions with the child. Family members will learn strategies to help the child eat enough at home and will address various issues concerning family relationships. Children will learn how to eat well on their own and will also discuss topics related to family dynamics. Participants assigned to the second group will receive 14 individual therapy sessions that will focus on the child and not include family members. Before each treatment session, parents will speak with the therapist to discuss progress and any new concerns or issues regarding the child's condition. The therapist will then work directly with the child to discuss what may be causing the child's signs of anorexia nervosa and how to handle difficult emotions associated with the disorder. Participants in both treatment groups will attend 1-hour therapy sessions that will occur weekly for 8 sessions, then biweekly for 4 sessions, and monthly for the last 2 sessions. Evaluations, lasting 3 to 4 hours, will occur before treatment begins, immediately following treatment, and 6 and 12 months post-treatment. Evaluations will consist of interviews and questionnaires used to assess whether treatment was effective in preventing participants from developing anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Living with family or guardian
* Medically stable for outpatient treatment
* Meets two to three criteria for anorexia nervosa
* Receiving a stable dose of psychotropic medication (if applicable)

Exclusion Criteria:

* Meets DSM-IV criteria for anorexia nervosa
* Current psychotic illness, alcohol or drug dependence, or medical or physical conditions known to influence eating, weight, or menstrual status
* Previous participation in study treatment
* Unable to withdraw from current psychological treatment

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2005-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Loeb, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Drury CR, Hail L, Rienecke RD, Accurso EC, Coelho JS, Lock J, Le Grange D, Loeb KL. Psychometric properties of the Parent Eating Disorder Examination Questionnaire. Int J Eat Disord. 2023 Sep;56(9):1730-1742. doi: 10.1002/eat.23999. Epub 2023 May 29. PMID 37248808
- [Derived] Loeb KL, Weissman RS, Marcus S, Pattanayak C, Hail L, Kung KC, Schron D, Zucker N, Le Grange D, Lock J, Newcorn JH, Taylor CB, Walsh BT. Family-Based Treatment for Anorexia Nervosa Symptoms in High-Risk Youth: A Partially-Randomized Preference-Design Study. Front Psychiatry. 2020 Jan 22;10:985. doi: 10.3389/fpsyt.2019.00985. eCollection 2019. PMID 32038326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period Oct 2007 to Feb 2011 primarily via physicians and other clinicians/centers evaluating or treating children and adolescents with eating disorder symptoms.
Groups:
- Family Based Therapy: Participants received family based therapy (FBT)
  Family-Based Therapy ("Maudsley Method"): The goal of FBT is to resolve the eating disorder and return the patient to healthy psychosocial and physiological development through active family involvement across three treatment phases. In Phase I, therapy is focused on the disordered eating. The therapist primarily makes careful, persistent requests for united parental action toward re-feeding and/or regulating eating habits and directs the discussion so as to create and reinforce a strong parental alliance around their efforts at feeding their child. In Phase II, the goal is to gradually transfer control over eating back to the participant, with the parents still maintaining general oversight and responsibility for continued progression toward healthy habits. In Phase III, the central goal is establishment of a healthy child or adolescent relationship with the parents where disordered eating is not the basis of interaction.
- Individual Supportive Psychotherapy: Participants received individual supportive psychotherapy (ISP)
  Individual Supportive Psychotherapy: The goal of ISP is for the patient to understand and address the psychological issues underlying the origin and maintenance of the eating disorder. This work is done directly with the child/adolescent. In this treatment, eating disorders are seen as complicated (e.g., they tend to mask other underlying difficulties). In Phase I, the aims are to establish a sound therapeutic relationship, obtain a comprehensive description of the eating problem and its development, identify underlying problems that might be responsible for the disordered eating, and inform the patient about the dangers of eating disorders. Phase II encourages participants to explore underlying emotional problems, facilitates self-disclosure and expression of feelings, and fosters independence. Phase III focuses on how other underlying issues might affect future adjustment.
Period: Overall Study
Arm/Group | Family Based Therapy | Individual Supportive Psychotherapy
Started | 43 | 16
Completed | 40 | 13
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Family Based Therapy: Participants received family based therapy (FBT)
- Individual Supportive Psychotherapy: Participants received individual supportive psychotherapy (ISP)
- Total: Total of all reporting groups
Arm/Group | Family Based Therapy | Individual Supportive Psychotherapy | Total
Number analyzed (Participants) | 43 | 16 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (2.0) | 14.8 (2.0) | 13.7 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 13 | 50
  Male | 6 | 3 | 9

OUTCOME MEASURES:

1. Secondary Outcome: Height
Description: This variable informs the calculation of the outcome variable of BMI Z-score.
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Family Based Therapy | Individual Supportive Psychotherapy
Number analyzed (Participants) | 40 | 13
inches | 61.3 (4.7) | 63.6 (4.1)

2. Secondary Outcome: Weight
Description: This variable informs the calculation of the outcome variable of BMI Z-score.
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Family Based Therapy | Individual Supportive Psychotherapy
Number analyzed (Participants) | 40 | 13
pounds | 94.9 (21.0) | 114.7 (29.1)

3. Secondary Outcome: BMI
Description: body mass index. This variable informs the calculation of the outcome variable of BMI Z-score.
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Family Based Therapy | Individual Supportive Psychotherapy
Number analyzed (Participants) | 40 | 13
kg/m^2 | 17.6 (2.0) | 19.7 (3.0)

4. Secondary Outcome: BMI Percentile
Description: Body Mass Index (BMI) percentile. This is not a primary outcome variable.
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Family Based Therapy | Individual Supportive Psychotherapy
Number analyzed (Participants) | 40 | 13
percentile | 30.1 (22.5) | 42.1 (29.4)

5. Primary Outcome: Body Mass Index (BMI) Z-score
Description: Z-score was calculated using the Baylor College of Medicine Children's Nutrition Research Center's online BMI calculator
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Family Based Therapy | Individual Supportive Psychotherapy
Number analyzed (Participants) | 40 | 13
z-score | -0.72 (.99) | -0.02 (.94)

ADVERSE EVENTS:
Arm/Group | Family Based Therapy | Individual Supportive Psychotherapy
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/16
Other Adverse Events (participants affected / at risk) | 0/43 | 0/16

LIMITATIONS AND CAVEATS:
Limitations include a small sample size and attrition leading to missing end-of-intervention data. In addition, participation with follow-up evaluations was poor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes